CLINICAL TRIAL: NCT01055067
Title: Multicenter Phase 2 Trial of ARQ 197 for Subjects With Relapsed or Refractory Germ Cell Tumors
Brief Title: ARQ 197 for Participants With Relapsed or Refractory Germ Cell Tumors
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was terminated early for futility according to the stopping rule of the Simon 2-stage design.
Sponsor: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ARQ197-A-U251
Record Dates: First submitted 2010-01-21; First posted 2010-01-25 (Estimated); Results first posted 2020-09-09 (Actual); Last update posted 2021-04-06 (Actual); Status verified 2021-03

CONDITIONS: Non-CNS Germ Cell Tumors (Seminomas and Nonseminomas)
MeSH Terms: conditions — Seminoma | interventions — ARQ 197

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Tivantinib (ARQ 197) (Experimental): 3 capsules of 120 mg each, administered twice a day (once in the morning and once in the evening - total daily dose of 720 mg) in continuous 4-week cycles
  Interventions: Drug: Tivantinib (ARQ 197)

INTERVENTIONS:
Drug: Tivantinib (ARQ 197) — Capsule, 120 mg, BID (360 mg), approximately 112 days
  Other Names: Tivantinib

SUMMARY:
This is a multicenter, single-arm study for safety and efficacy.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically-confirmed non-central nervous system germ cell tumor (non-CNS GCT), both seminomas and nonseminomas are allowed.
2. Male subjects 16 years of age or older.
3. Eastern Cooperative Oncology Group (ECOG) performance status of equal to or less than 1.
4. Documented progression during or following equal to or greater than 1 prior platinum-containing chemotherapy regimen(s) (no limit to number of lines of prior treatment), and considered platinum-resistant by the Investigator. Subjects who have progressed or whose tumors have recurred after stem cell transplantation are also allowed.
5. All subjects must have either declined or not be a candidate for curative therapy. In general, this means a subject would have to have progressive disease (PD) after receiving high-dose chemotherapy, have certain features making them ineligible for high-dose chemotherapy, or have refused high-dose chemotherapy despite being informed of its curative potential.
6. Subjects must have radiographically measurable disease as defined by RECIST 1.1 and meet one of the following criteria:

   * Documented germ cell tumor progression based on radiographic measurements;
   * Elevated serum tumor markers in case of radiographically measured stable disease.
7. Subjects should be able to provide written informed consent, comply with protocol visits and procedures, be able to take oral medication, and not have any active infection or chronic co-morbidity that would interfere with therapy.
8. Subjects must agree to use double-barrier contraceptive measures or avoidance of intercourse during the study and for 90 days after the last dose of study drug.
9. Adequate bone marrow, liver, and renal functions, defined as:

   * Platelet count equal to or greater than 75 times 10^9/L;
   * Hemoglobin equal to or greater than 9.0 g/dL;
   * Absolute neutrophil count (ANC) equal to or greater than 1.5 times 10^9/L;
   * Total bilirubin equal to or less than 2.5 mg/dL;
   * Alanine aminotransaminase (ALT) and aspartate aminotransaminase (AST) equal to or less than 2.5 times the upper limit of normal (ULN) (equal to or less than 5 times the ULN for subjects with liver metastases);
   * Serum creatinine equal to or less than 1.5 times the ULN.
10. Subjects must be fully informed about their illness and the investigational nature of the study protocol (including foreseeable risks and possible side effects) and must sign and date an Independent Ethics Committee or Institutional Review Board approved informed consent form (including Health Insurance Portability and Accountability Act authorization, if applicable) before performance of any study specific procedures or tests.

Exclusion Criteria:

1. Previous or concurrent cancer that is distinct from GCT in primary site or histology, EXCEPT treated basal cell carcinoma, superficial bladder tumors (Ta, Tis & T1). Any cancer curatively treated equal to or greater than 3 years prior to enrollment is permitted.
2. History of cardiac disease:

   * Congestive heart failure defined as Class II to IV per New York Heart Association classification.
   * Active coronary artery disease.
   * Previously diagnosed bradycardia or other cardiac arrhythmia defined as equal to or greater than Grade 2 according to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE), version 4.0, or uncontrolled hypertension.
   * Myocardial infarction that occurred within 6 months prior to study entry (myocardial infarction that occurred greater than 6 months prior to study entry is permitted).
3. Active clinically serious infection(s) defined as equal to or greater than Grade 2 according to NCI CTCAE, version 4.0.
4. Known metastatic brain or meningeal tumors, unless the subject is greater than 6 months from definitive therapy, has a negative imaging study within 4 weeks of first dose of study drug and is clinically stable (no concomitant therapy, including supportive therapy with steroids or anticonvulsant medications) with respect to the tumor at the time of first dose of study drug.
5. Any primary CNS GCT.
6. Concurrent treatment with anticancer therapies including cytotoxic chemotherapy, immunotherapy, radiotherapy, vaccines or investigational therapy during the study or within 3 weeks of first dose of study drug.
7. Any major surgical procedure within 3 weeks prior to first dose of study drug.
8. Prior therapy with c-MET inhibitors, including ARQ197.
9. Substance abuse or medical, psychological or social conditions that may, in the opinion of the Investigator, interfere with the subject's participation in the clinical study or evaluation of the clinical study results.
10. Any condition that is unstable or that could jeopardize the safety of the subject and the subject's protocol compliance, including known human immunodeficiency virus, hepatitis B virus or hepatitis C virus infection.
11. Inability to swallow oral medications.

Min Age: 16 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2010-02-02 (Actual); Primary Completion 2011-11-30 (Actual); Study Completion 2011-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Study Leader, Study Director — Daiichi Sankyo
Locations (10):
- United States (6):
  - Los Angeles, California
  - Orlando, Florida
  - Indianapolis, Indiana
  - St Louis, Missouri
  - New York, New York
  - Philadelphia, Pennsylvania
- France (2):
  - Lyon
  - Villejuif
- United Kingdom (2):
  - Leeds
  - London

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 27 participants who met all inclusion and no exclusion criteria were enrolled and treated at 7 clinic sites in the United States, 2 in France, and 2 in the United Kingdom. Of the 27 enrolled, 21 were included in Stage 1 in which the interim futility analysis was performed per the Simon 2-stage design.
Pre-assignment Details: Based on the Simon 2-stage design, 21 participants were enrolled (Stage 1). If <2 had either a complete response (CR) or partial response (PR), then the study was terminated. If ≥2 had either CR or PR, then enrollment was extended to 41 participants. After Stage 2 with 41 participants, treatment was effective if ≥5 had CR or PR after 4 cycles.
Groups:
- Total: All enrolled participants who received at least 1 dose of study drug in the study.
Period: Overall Study
Arm/Group | Total
Started | 27
Completed (Defined as participants who had progressive disease) | 27
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Demographic and baseline characteristics were assessed in the Full Analysis Set.
Arm/Group | Total
Number analyzed (Participants) | 27
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 27
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.0 (11.59)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 27
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 23
  Other | 4

OUTCOME MEASURES:

1. Primary Outcome: Best Overall Response and Objective Response Rate Following Treatment With Tivantinib (ARQ 197) in Participants With Relapsed or Refractory Germ Cell Tumors
Description: The best overall response was the best response (in the order of confirmed complete response [CR], confirmed partial response [PR], unconfirmed CR, unconfirmed PR, stable disease [SD], and progressive disease [PD]) among all overall responses recorded from the start of treatment until the participant withdrew from the study. Objective response was defined as the number of participants with confirmed CR and confirmed PR after 4 cycles of therapy with ARQ 197. According to Response Evaluation Criteria in Solid Tumors v 1.1, CR was defined as a disappearance of all target lesions, PR was defined as at least a 30% decrease in the sum of diameters of target lesions, and SD was defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, defined as at least a 20% increase in the sum of diameters of target lesions.
Time Frame: Baseline up to first objective response, up to 1 year 9 months postdose
Population: Objective response rate was assessed in the Full Analysis Set.
Measure: Count of Participants; unit: Participants
Groups:
- Stage 1: ARQ 197 360 mg BID: Participants who were enrolled in Stage 1 of the Simon 2-stage design and received ARQ 197 360 mg twice a day (BID) (with a 720 mg total daily dose) in participants with relapsed or refractory non-central nervous system germ cell tumor (non-CNS GCT).
Arm/Group | Stage 1: ARQ 197 360 mg BID | Total
Number analyzed (Participants) | 21 | 27
Participants
  Confirmed CR | 0 | 0
  Confirmed PR | 0 | 0
  Stable disease | 3 | 5
  Progressive disease | 16 | 20
  Objective response rate | 0 | 0

2. Secondary Outcome: Progression-Free Survival Following Treatment With Tivantinib (ARQ 197) in Participants With Relapsed or Refractory Germ Cell Tumors
Description: Progression-free survival (PFS) is defined as the time from the date of the start of study treatment to the earlier of the dates of the first documentation of progressive disease (PD) or death due to any cause. According to Response Evaluation Criteria in Solid Tumors v 1.1, progressive disease was defined as at least a 20% increase in the sum of diameters of target lesions.
Time Frame: Baseline up to progressive disease or death (whichever occurs first), up to 1 year 9 months postdose
Population: Progression-free survival was assessed in the Full Analysis Set.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Stage 1: ARQ 197 360 mg BID | Total
Number analyzed (Participants) | 21 | 27
weeks | 4.3 [4.1 to 8.0] | 4.3 [4.1 to 8.0]

3. Secondary Outcome: Overall Survival Following Treatment With Tivantinib (ARQ 197) in Participants With Relapsed or Refractory Germ Cell Tumors
Description: Overall survival (OS) was defined as the time from the date of the start of study treatment to the date of death due to any cause.
Time Frame: Baseline up to death (any cause), up to 1 year 9 months postdose
Population: Overall survival was assessed in the Full Analysis Set.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Stage 1: ARQ 197 360 mg BID | Total
Number analyzed (Participants) | 21 | 27
months | 6.2 [3.5 to 7.7] | 5.9 [3.5 to 7.7]

4. Secondary Outcome: Treatment-Emergent Adverse Events Reported in ≥ 10% of Participants Following Treatment With Tivantinib (ARQ 197) in Participants With Relapsed or Refractory Germ Cell Tumors
Description: Treatment-emergent adverse events (TEAEs) were defined as an adverse event (AE) that occurs, having been absent before the first dose of study drug, or has worsened in severity or seriousness after the first dose until 30 days after the last dose.
Time Frame: Baseline up to 30 days after last dose, up to 1 year 9 months postdose
Population: Adverse events were assessed in the Safety Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | Stage 1: ARQ 197 360 mg BID | Total
Number analyzed (Participants) | 21 | 27
Participants
  Any TEAEs | 19 | 25
  Gastrointestinal Disorders | 8 | 11
  Constipation | 2 | 3
  Nausea | 6 | 7
  Vomiting | 4 | 4
  General Disorders & Administration Site Conditions | 12 | 15
  Fatigue | 7 | 10
  Edema peripheral | 3 | 4
  Metabolism and Nutrition Disorders | 3 | 6
  Decreased appetite | 3 | 4
  Musculoskeletal and Connective Tissue Disorders | 4 | 6
  Back pain | 2 | 3
  Nervous System Disorders | 7 | 11
  Neuropathy peripheral | 3 | 3
  Respiratory, Mediastinal, and Thoracic Disorders | 8 | 12
  Cough | 3 | 6
  Dyspnea | 4 | 6

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events (TEAEs) were collected from baseline up to 30 days after last dose, up to 1 year 9 months.
Description: Treatment-emergent adverse events (TEAEs) were defined as an adverse event (AE) that occurs, having been absent before the first dose of study drug, or has worsened in severity or seriousness after the first dose until 30 days after the last dose.
Arm/Group | Stage 1: ARQ 197 360 mg BID | Total
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/27
Serious Adverse Events (participants affected / at risk) | 6/21 | 9/27
Other Adverse Events (participants affected / at risk) | 11/21 | 15/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Stage 1: ARQ 197 360 mg BID (N=21) | Total (N=27)
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Vision blurred (Eye disorders) | 1 | 1
Peritoneal haemorrhage (Gastrointestinal disorders) | 0 | 1
Hypersensitivity (Immune system disorders) | 1 | 1
Cellulitis (Infections and infestations) | 1 | 1
Pneumonia (Infections and infestations) | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Cerebral haemorrhage (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 1 | 1
Sciatica (Nervous system disorders) | 0 | 1
Spinal cord compression (Nervous system disorders) | 1 | 1
Superior vena caval occlusion (Vascular disorders) | 1 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Stage 1: ARQ 197 360 mg BID (N=21) | Total (N=27)
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 2
Dry mouth (Gastrointestinal disorders) | 1 | 1
Nausea (Gastrointestinal disorders) | 3 | 4
Vomiting (Gastrointestinal disorders) | 2 | 2
Fatigue (General disorders) | 5 | 7
Pneumonia (Infections and infestations) | 1 | 1
Decreased appetite (Metabolism and nutrition disorders) | 2 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Dysgeusia (Nervous system disorders) | 1 | 1
Syncope (Nervous system disorders) | 1 | 1
Insomnia (Psychiatric disorders) | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 1

LIMITATIONS AND CAVEATS:
The study was terminated early for futility according to the stopping rule of the Simon 2-stage design since no participants in Stage 1 had achieved either a complete response or partial response. Enrollment halted and Stage 2 did not occur.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No